CLINICAL TRIAL: NCT00208039
Title: Pilot Trial of Surfactant Booster Prophylaxis For Ventilated Preterm Neonates Less Than or Equal to 1250 gm Birthweight Ver 4.0
Brief Title: Pilot Trial of Surfactant Booster Prophylaxis For Ventilated Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Women & Children's Hospital of Buffalo (Other); Children's Mercy Hospital Kansas City (Other); St. Louis Children's Hospital (Other); UCSF Benioff Children's Hospital Oakland (Other); Alta Bates Summit Medical Center (Other); Long Island Jewish Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-9-3983
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Respiratory Distress Syndrome; Bronchopulmonary Dysplasia
Keywords: Prematurity; Lung Disease; Hyaline Membrane; Surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia; Premature Birth; Lung Diseases | interventions — calfactant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Infasurf — Infasurf 3 cc/kg instilled via endotracheal tube, repeated 3 and 7 days later if infant stable and continues to meet criteria
  Other Names: Infasurf (calfactant, manufactured for INOTherapeutics, Clinton NJ by ONY Inc., Amherst, NY)

SUMMARY:
A research study that will evaluate if giving surfactant medication to premature babies weighing < 1250 gm at birth during the second and third weeks of life will help their lungs. We are enrolling those premature babies who continue to require the breathing tube and the mechanical ventilator at days 7-10 of life.

DETAILED DESCRIPTION:
Pulmonary surfactant is required for normal lung function. Data from a previous study suggest that as many as 75% of chronically ventilated extremely low birthweight premature infants have at least one episode of surfactant dysfunction beyond the first week of life, as measured in vitro, associated with a low surfactant protein B content. Furthermore, episodes of surfactant dysfunction are significantly associated with clinically significant respiratory decompensations. We hypothesize that booster doses of surfactant given during the second and third week of life to extremely low birth weight premature infants requiring persistent intubation and mechanical ventilation will improve their respiratory status during the first 28 days of life. We propose to enroll premature infants < 1250 gm birthweight, between days 7 and 10 of life who are intubated, and mechanically ventilated. Infants requiring persistent intubation and mechanical ventilation for respiratory support at 7-10 days of life will receive a total of 3 doses of Infasurf surfactant, 3 days apart, at the standard dose of 3 ml/kg. Primary outcome is the change in area under the respiratory severity score curve between days 7 and 28 of life. Total sample size is 88 infants, study duration is 36 months, and recruitment of study patients will occur at The Hospital of the University of Pennsylvania, in Philadelphia PA, Women and Children's Hospital in Buffalo, St. Louis Children's Hospital in St. Louis MO, Mercy Children's Hospital in Kansas City, Oakland Children's and Alta Bates Medical Center in Berkeley, CA and Long Island Jewish Medical Center, NY.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to1250 gm birthweight
* Day 7-10 of life
* Intubated and mechanically ventilated at day 7-10 of life

Exclusion Criteria:

* Infants intubated solely for apnea
* Serious congenital malformations
* Life expectancy < 7 days from enrollment
* Pulmonary hemorrhage at time of enrollment
* Active air leak syndrome at time of enrollment
* Bilateral grade IV intracranial hemorrhage
* Postnatal systemic steroid therapy for lung disease

Note: Prior surfactant therapy at birth is neither an inclusion nor exclusion criterion.

Ages: 7 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2004-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Surfactant therapy will decrease the mean area under the curve(of the plots of daily respiratory severity scores between days 7 and 28 of life), by 33% from historic controls. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Posencheg, MD, Principal Investigator — University of Pennsylvania/Children's Hospital of Philadelphia; Roberta A Ballard, MD, Principal Investigator — University of California, San Francisco Medical Center

REFERENCES:
- [Background] Merrill JD, Ballard RA, Cnaan A, Hibbs AM, Godinez RI, Godinez MH, Truog WE, Ballard PL. Dysfunction of pulmonary surfactant in chronically ventilated premature infants. Pediatr Res. 2004 Dec;56(6):918-26. doi: 10.1203/01.PDR.0000145565.45490.D9. Epub 2004 Oct 20. PMID 15496605